CLINICAL TRIAL: NCT01086189
Title: Does Green Tea Affect Postprandial Glucose, Insulin and Satiety in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Other Study IDs: 2009/66
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
Green tea consumption could lower the risk of type II diabetes, as suggested by epidemiological studies. There is also evidence from intervention studies that green tea can decrease blood glucose levels and contribute to weight loss.

The aim with this study is therefore to examine the postprandial effects of green tea on glycemic index, insulin levels and satiety in healthy individuals after the consumption of a meal.

DETAILED DESCRIPTION:
The study was conducted on 14 healthy volunteers, with a crossover design. Participants were randomized to either green tea or water. This was consumed together with a breakfast consisting of white bread. Blood samples were drawn at 0, 15, 30, 45, 60, 90 and 120 minutes. Participants completed two different satiety scores at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 14 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-12; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose and insulin

SECONDARY OUTCOMES:
Postprandial satiety

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Josic J, Olsson AT, Wickeberg J, Lindstedt S, Hlebowicz J. Does green tea affect postprandial glucose, insulin and satiety in healthy subjects: a randomized controlled trial. Nutr J. 2010 Nov 30;9:63. doi: 10.1186/1475-2891-9-63. PMID 21118565